CLINICAL TRIAL: NCT06964659
Title: Sulforaphane-Smart® on Lipid and Glucose Metabolism, Inflammation, Adiposity and Microbiome of Overweight Adults "SANO"
Brief Title: Chronic Intervention With Sulforaphane-Smart® in Overweight and Obese Adults
Acronym: SANO-Chronic
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mª Jesús Periago (Other)
Collaborators: Ingredalia Company (Unknown); Spanish National Research Council (CEBAS-CSIC) (Unknown)
Responsible Party: Sponsor-Investigator, Mª Jesús Periago, PhD Full Professor of Food Science and Nutrition, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SANO Project (Chronic); CPP2022-009528 (Other: Ministerio de Ciencia, Innovación y Universidades)
Record Dates: First submitted 2025-03-07; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Overweight
Keywords: Glucosinolates; Isothiocyanates; Sulforaphane; Gut microbiota; Inflammation; Oxidative stress
MeSH Terms: conditions — Obesity; Overweight; Inflammation | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The volunteers will be randomly assigned to the intervention groups. The experimental group (with 20 volunteers) intake daily the Sulforaphane-Smart® pill during 12 weeks, and the placebo group (with 20 volunteers) intake the placebo pill in parallel during the same period.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulforaphan-Smart® formula (Experimental): The volunteers of the experimental group will intake of Sulforaphan-Smart® formula to evaluate if the chronic consumption of GSL/ITC, during the intervention period of 12 weeks, could modulate the glucidic and lipid metabolism, the biomarkers related to chronic inflammation and oxidative stress and the gut microbiota in overweight and obese volunteers.
  Interventions: Dietary Supplement: Sulforaphan-Smart® formula
- Control/Placebo (Placebo Comparator): The volunteers of placebo group will intake the placebo formula or pill to objectively separate the effects of the drug under study (Sulforaphane Smart® formula) during the intervention period of 12 weeks.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Dietary Supplement: Sulforaphan-Smart® formula — Volunteers will intake a daily dose of Sulforaphan-Smart® pill for 12 weeks (84 days)
  Other Names: GLS/ITC group
  Arms: Sulforaphan-Smart® formula
Other: Control (placebo) group — Volunteers will intake a daily dose of placebo pill for 12 weeks (84 days)
  Other Names: PL group
  Arms: Control/Placebo

SUMMARY:
The Sulforaphane-Smart® formula is a pill, patented by the company INGREDALIA, prepared with broccoli by-products which have been concentrated and enriched in glucosinolates/isothiocyanates (GLS/ITCs).

The goal of this intervention study is to evaluate if the chronic consumption of GSL/ITC (Sulforaphane Smart® formula) could modulate the biomarkers related to chronic inflammation, oxidative stress and gut microbiota in overweight and obese volunteers.

In order to reach this goal, the volunteers will take daily the Sulforaphane Smart® formula during 12 weeks (total of 84 days). Anthropometric measurements will be taken and biological samples of blood, urine and feces will be collected at the beginning of the intervention (initial time), after six weeks of the intervention (Time 6 weeks) and at the end of the intervention (Time 12 weeks).

DETAILED DESCRIPTION:
Sulforaphan-Smart® is formula patented by the company INGREDALA (patented by INGREDALIA: EP3123874B1). This clinical trial will provide information about the beneficial effects of the consumption of Sulforaphan Smart® on glucidic and lipid metabolism, inflammation, adiposity, antioxidant status and microbiome of adults with overweight or obesity.

The study will be conducted with a total of 40 adults with overweight and obesity (BMI 25 to 34.9 Kg/m2) from both sexes. Volunteers will be divided into two groups according to the randomized-controlled and parallel design protocol, with two arms (experimental and placebo groups) with 20 volunteers per group.

During 12 weeks the experimental group will intake one daily dose of Sulforaphan Smart®, meanwhile the placebo group will intake one daily dose of placebo. Biological samples (blood, urine and feces) will be taken during the intervention and the following experimental parameters will be taken at the beginning (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks):

* Anthropometric study will be performed with a Tanita Body Weight Scale (DC-430MAP).
* Biochemical parameters of plasma related to glucidic and lipid metabolism.
* Analysis of Biomarkers of inflammation in plasma (C-reactive protein, adiponectin, IL-6, IL-1β and IL-8).
* Analysis of oxidative stress biomarkers in plasma and urine: determination of isoprostanes and malonaldehyde concentrations.
* Analysis of fecal microbiota by 16SrRNA sequencing after extraction of total DNA from feces.
* Analysis of Short Chain Fatty Acids by GLC in feces as metabolites of the fecal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* BMI: overweight and obese (BMI 25-34,9 Kg/m2)
* No digestive or intestinal diseases
* Age between 20 and 45 years old
* Not having antibiotics during the previous three months
* Not having pharmacological treatment
* Not being smokers
* Not following restrictive diets (vegetarian/vegan diet) or nutritional supplement

Exclusion Criteria:

* BMI: low and normal weight
* Age different from that required
* Digestive or intestinal diseases
* Having antibiotics during the previous three months
* Having pharmacological treatments
* Following restrictive diets (vegetarian/vegan diet) or nutritional supplement
* Smoker

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the concentration of plasmatic glucose | Plasmatic glucose concentration will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  Glucose concentration will be analyzed in plasma samples of both experimental and placebo groups, to determine the effect of the daily intake of Sulforaphan-Smart® formula.
Changes in the concentration of plasmatic insulin | Plasmatic insulin concentration will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  Insulin concentration will be analyzed in the plasma samples in both experimental and placebo groups, to determine the effect of the daily intake of Sulforaphan-Smart® forrmula.
Changes in the HOMA-IR | HOMA-IR index will be calculated at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  The HOMA-IR index will be calculated using the plasmatic concentration of glucose and insulin, to determine the insulin resistance index in both experimental and placebo groups after the daily intake of Sulforaphan-Smart® formula.
Changes in the concentration of lipid metabolism parameters of plasma | Lipid metabolism parameters will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  Lipid metabolism parameters of plasma including total cholesterol, LDL-C, HDL-C and triglycerides will be analyzed in the plasma samples in both experimental and placebo groups, to determine the effect of the daily intake of Sulforaphan-Smart® formula.
Changes of C-reactive protein in plasma | C-reactive protein will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  The concentration of C-reactive protein will be analyzed, in plasma samples in both experimental and placebo groups as biomarker of inflammation, to evaluate the effect of the daily consumption of Sulforaphan-Smart®. The concentration of this biomarker will be analyzed using an ELISA kit, following the manufacturer's instructions.
Changes of TNF-α in plasma | TNF-α will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  Tumor Necrosis Factor alfa (TNF-α) will be determined in samples, of both experimental and placebo groups, to determine the effect of the daily consumption of Sulforaphan-Smart® in chronic inflammation. The concentration of this biomarker will be analyzed using an ELISA kit, following the manufacturer's instructions.
Changes of Interleukins in plasma | Interleukins will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of intervention (Time 12 weeks).
  Interleukins (IL-6, IL-1β and IL-8) will be analysed in samples of both experimental and placebo groups, to evaluate the effect of the daily consumption of Sulforaphan-Smart® on chronic inflammation. The concentration of these biomarkers will be analyzed using an ELISA kit, following the manufacturer's instructions.
Changes of MDA in plasma | MDA will be analysed at the beginning of the intervention (initial time), at six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  Malonaldehyde (MDA) will be analysed in plasma samples of bth experimental and placebo groups to evaluate the effect of the daily consumption of Sulforaphan-Smart® formula on the oxidative stress. For this purpose MDA concentration will be analysed in plasma samples using an ELISA kit, following the manufacturer's instructions.
Changes of isoprostanes concentration in urine | Isosprotanes concentration will be analysed in urine at the beginning of the intervention (initial time), at six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  Isoprostanes concentration will be analysed in urine samples of both experimental and placebo groups , with the aim to evaluate the effect of the daily consumption of Sulforaphan-Smart® formula on oxidative stress. This biomarker will be analysed using an ELISA kit, following the manufacturer's instructions
Changes of MDA concentration in urine | MDA concentration will be analysed at the beginning of the intervention (initial time), at six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  Malonaldehyde (MDA) concentration will be analysed in urine samples of both experimental and placebo groups, with the aim to evaluate the effect of the daily consumption of Sulforaphan-Smart® formula on oxidative stress. The concentration of this biomarker will be determined using an ELISA kit, following the manufacturer's instructions.
Changes in microbiota | The composition of the gut microbiota will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The effect of the daily intake of Sulforaphan-Smart® formula on gut microbiota will be determined by 16S rRNA sequencing, after the extraction of total faecal DNA.
Changes of SCFAs in feces | The concentration of SCFAs in feces will be analysed at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The changes in the concentration of short-chain fatty acids (SCFAs) in feces after the daily intake of Sulforaphan-Smart® formula will be analysed by gas chromatography (GC-FID).

SECONDARY OUTCOMES:
Changes in the body mass index | BMI will be taken at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The measurement of the body mass index (BMI) will be carried out throughout the intervention study, in both experimental and placebo groups. For this purpose, weight (kg) and height (cm) will be registered and used to calculate the total BMI (kg/m^2).
Changes in the waist-to-hip ratio | The WHR will be measured at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The measurements of the waist-to-hip ratio (WHR) will be carried out throughout the intervention study, in both experimental and placebo groups. The circumference of the waist and hip will be registered (cm) and used to calculate the WHR.
Changes in body fat mass percentage | Fat mass percentage will be registered at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The fat mass percentage will measure using a Tanita DC-430MAP body scale, in both experimental and placebo groups, to determine possible changes after the daily intake of Sulforaphane Smart® formula.
Changes in body fat free mass percentage | Fat free mass percentage will be registered at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The fat free mass percentage will measure with a Tanita DC-430MAP body scale in both experimental and placebo groups, to determine possible changes after the daily intake of Sulforaphane Smart® formula.
Changes in body water percentage | Body water percentage will be registered at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The body water percentage will measure with a Tanita DC-430MAP body scale in both experimental and placebo groups, to determine possible changes after the daily intake of Sulforaphane Smart® formula.
Changes in body bone mass percentage | Body bone mass percentage will be registered at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The body bone mass percentage will measure with a Tanita DC-430MAP body scale, in both experimental and placebo groups, to determine possible changes after the daily intake of Sulforaphane Smart® formula.
Changes in visceral fat index | Visceral fat index will be registered at the beginning of the intervention (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  The visceral fat index will measure with a Tanita DC-430MAP body scale, in both experimental and placebo groups, to determine possible changes after the daily intake of Sulforaphane Smart® formula.
Evaluation of food intake questionnaire | The 24-hours food intake questionnaire will be registered at the beginning (initial time), after six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks)
  The volunteers will provide information about the 24-hours food intake questionaries before the collection of the biological samples, to quantify the intake on nutrients and energy.
Evaluation of the dietary habits | Mediterranean Diet Adherence Questionnaire will be completed at the beginning of the intervention (initial time), at six weeks (Time 6 weeks) and at the end of the intervention (Time 12 weeks).
  All volunteers will fill a "Mediterranean Diet adherence" questionnaire to evaluate the adherence of the diet profile.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío González Barrio, PhD, Principal Investigator — Universidad de Murcia; María Jesús Periago Castón, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Edificio Pleyades-Vitalys 5ª y 6ª planta, Campus Universitario, Espinardo, Murcia, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: A systematic review about the nutritional interest of glucosinolates, including human intervention studies — https://doi.org/10.3389/fnut.2021.648788